CLINICAL TRIAL: NCT02134691
Title: Randomized Trial of Prolonged Exposure for the Treatment of Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mildred Vera, Professor, University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SC1MH090599 (NIH)
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder (PTSD); Prolonged Exposure (PE)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Exposure (Experimental): Behavioral: Prolonged Exposure (PE) PE is a 16 week, 90 minute culturally informed treatment program.
  Interventions: Behavioral: Prolonged Exposure
- Applied Relaxation (Active Comparator): Behavioral: Applied Relaxation (AR) AR is a 16 week, 90 minute treatment program.
  Interventions: Behavioral: Applied Relaxation

INTERVENTIONS:
Behavioral: Prolonged Exposure
  Arms: Prolonged Exposure
Behavioral: Applied Relaxation
  Arms: Applied Relaxation

SUMMARY:
This project will examine the impact of PE therapy for the treatment of PTSD with a sample of Latinos. The need to provide effective treatment to Spanish-speaking Latinos with PTSD is critical given the high prevalence of PTSD among Latinos. Furthermore, PTSD remains an under detected and under treated condition. Untreated PTSD has a substantial impact on health, functioning and quality of life. PE is one of the most empirically supported psychological interventions for PTSD. However, most studies that evidence the efficacy of PE have been conducted mainly with English-speaking Caucasian populations. This study has the potential to contribute to improvements in the well-being of Spanish-speaking Latinos with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* 18 to < 65 years
* Meet diagnostic criteria for PTSD
* Spanish speaker
* Allow recording of assessments and therapy

Exclusion Criteria:

* Significant current suicidal or homicidal ideation
* History of bipolar, schizophrenia or psychotic disorder
* Alcohol or drug abuse during the past three months
* Current high risk of being assaulted (i.e., living with domestic violence)
* Current psychotherapy to treat PTSD
* Unable to provide informed consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2013-08; Primary Completion 2018-06-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Clinician Administered PTSD Scales (CAPS) | 6 months

SECONDARY OUTCOMES:
Change in SF-12 | 6 months
Change in Sheehan Disability Scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mildred Vera, Ph.D, Principal Investigator — University of Puerto Rico Medical Sciences Campus
Locations (1):
- University of Puerto Rico, Medical Sciences Campus, San Juan, Puerto Rico